CLINICAL TRIAL: NCT05681728
Title: A Phase II Study Evaluating the Efficacy and Safety of Pembrolizumab in Combination With Chemotherapy as Neoadjuvant Therapy for Triple-negative Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Ma Fei，MD, Deputy Director of the Department of Medical Oncology, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC3340
Record Dates: First submitted 2022-12-28; First posted 2023-01-12 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2022-12

CONDITIONS: Breast Cancer
Keywords: breast cancer; neoadjuvant therapy; immunotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — pembrolizumab; Paclitaxel; Epirubicin; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab combined with chemotherapy (Experimental)
  Interventions: Drug: Pembrolizumab; Drug: Paclitaxel; Drug: Epirubicin; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Pembrolizumab — On Day 1 of each cycle in the neoadjuvant and adjuvant phases of the study for a total of 17 cycles; intravenous (IV) infusion
Drug: Paclitaxel — On Day 1 of Cycles 1-4 in the neoadjuvant phase of the study; IV infusion
Drug: Epirubicin — On Day 1 of Cycles 5-8 of the neoadjuvant phase of the study; IV injection
Drug: Cyclophosphamide — On Day 1 of Cycles 5-8 of the neoadjuvant phase of the study; IV infusion

SUMMARY:
A Phase II study that evaluating the efficacy and safety of pembrolizumab in combination with chemotherapy as neoadjuvant therapy for triple-negative breast cancer in the Chinese population

ELIGIBILITY:
Inclusion Criteria:

Men or women who are 18 years of age or older on the date of signing the informed consent form.

Pathologically confirmed invasive ductal carcinoma of the breast with stage T1c and N 1-3, or cT2-T4/N0-3.

Patients with triple-negative breast cancer according to the most recent American Society of Clinical Oncology/American College of Pathologists guidelines.

Has Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 performed within 10 days of treatment initiation.

Female subjects were not pregnant, breastfeeding, and had been on birth control for at least 24 months after the last dose.

Subjects can sign informed consent to participate in the study. Appropriate organ function; All screening period laboratory tests should be completed within 10 days prior to the start of study therapy.

Exclusion Criteria:

Has a history of invasive malignancy ≤5 years prior to signing informed consent except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer.

Has received prior chemotherapy, targeted therapy, and radiation therapy within the past 12 months.

Has received prior therapy with an anti-programmed cell death protein 1 (anti-PD-1), anti-programmed death - ligand 1 (anti-PD-L1), or anti-PD-L2 agent or with an agent directed to another co-inhibitory T-cell receptor (e.g., cytotoxic T-lymphocyte-associated antigen-4 [CTLA-4], OX-40, CD137 [tumor necrosis factor receptor superfamily member 9 (TNFRSF9)]) or has previously participated in a pembrolizumab (MK-3475) clinical study.

Is currently participating in or has participated in an interventional clinical study with an investigational compound or device within 4 weeks of the first dose of treatment in this current study.

Has received a live vaccine within 30 days of the first dose of study treatment.

Has an active autoimmune disease that has required systemic treatment in past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs).

Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy (i.e., dosing exceeding 10 mg daily of prednisone or equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment.

Has a known history of Human Immunodeficiency Virus (HIV). Has known active Hepatitis B or Hepatitis C. Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.

Has an active infection requiring systemic therapy. Has significant cardiovascular disease, such as: history of myocardial infarction, acute coronary syndrome or coronary angioplasty/stenting/bypass grafting within the last 6 months OR congestive heart failure (CHF) New York Heart Association (NYHA) Class II-IV or history of CHF NYHA Class III or IV.

Is pregnant or breastfeeding, or expecting to conceive children within the projected duration of the study, starting with the screening visit through 12 months after the last dose of study treatment for participants who have received cyclophosphamide, and for 6 months after the last dose of study treatment for participants who have not.

Has a known hypersensitivity to the components of the study treatment or its analogs.

Has a known history of active tuberculosis (TB, Bacillus Tuberculosis).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate using the definition of ypT0/Tis ypN0 (i.e., no invasive residual in breast or nodes; noninvasive breast residuals allowed) at the time of definitive surgery | Up to approximately 27-30 weeks
  pCR rate (ypT0/Tis ypN0) is defined as the percentage of participants without residual invasive cancer on hematoxylin and eosin evaluation of the complete resected breast specimen and all sampled regional lymph nodes following completion of neoadjuvant systemic therapy by current American Joint Committee on Cancer (AJCC) staging criteria assessed by the local pathologist at the time of definitive surgery.

SECONDARY OUTCOMES:
Event-free Survival (EFS) as assessed by Investigator | Up to approximately 8 years
  EFS is defined as the time from randomization to any of the following events: progression of disease that precludes surgery, local or distant recurrence, second primary malignancy (breast or other cancers) or death due to any cause
Percentage of participants who experience an adverse event (AE) | Up to approximately 52 weeks
  An AE is defined as any untoward medical occurrence in a participant administered study treatment which does not necessarily have to have a causal relationship with this treatment. An AE can be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of study treatment or protocol-specified procedure, whether or not considered related to study treatment or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a pre-existing condition that is temporally associated with the use of study treatment, is also an AE

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No